CLINICAL TRIAL: NCT03683004
Title: Chemotherapy-Related Changes in Neurocognitive Function and Symptoms in Colorectal Cancer Patients: A Pilot Study
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0228-17-EP
Record Dates: First submitted 2018-07-05; First posted 2018-09-25 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CRC patients (Ctx+ group): Postoperative CRC patients scheduled to begin CTX
- CRC patients (CT- group): Postoperative CRC patients who do not receive CTX
- Healthy control group: Study participants that are demographically matched to CRC study patients and meet all inclusion criteria

SUMMARY:
Cancer treatments have successfully improved cancer outcomes but frequently negatively impact quality of life in cancer survivors. In particular, chemotherapy (CTX) has been associated with impaired cognitive abilities such as concentration and memory. The goal is to investigate the neural mechanisms of chemotherapy-related cognitive impairment (CRCI) using an interdisciplinary translational approach. Previous research in this area lacks diversity in studied cancer populations and treatments focusing primarily on breast cancer and provides limited understanding of how CRCI emerges from changes in neural structure, function, and connectivity. To overcome these limitations, this feasibility/pilot study aims to investigate CRCI in patients with colorectal cancer (CRC).

DETAILED DESCRIPTION:
A growing public health and oncology nursing concern is the likelihood of colorectal cancer (CRC) survivors experiencing decline in long-term physical and mental functional status following cancer diagnosis and treatment. Prior to receiving treatment, cognitive impairment in processing speed, spatial working memory, and verbal memory has been noted in 45% of CRC patients relative to 15% of healthy controls (HC). Following adjuvant chemotherapy, cognitive function is more impaired in CRC patients who received chemotherapy (Ctx+ group) compared to CRC patients not receiving chemotherapy (Ctx- group) and HC participants. These studies show: (1) CRC patients are at a high risk for cognitive impairment and (2) Ctx+ patients are more likely to decline in cognitive function during treatment. These cancer and chemotherapy-related changes in cognitive function have been associated with several quality of life factors, including physiological and concurrent symptoms, and physical and mental functional status. In contrast, the neural mechanisms of cognitive impairment in CRC patients is related to changes in the Executive Function Network (EFN). The EFN promotes long-range communication between frontal and parietal cortical regions, and is associated with attentional control processes. The empirical goals studying CRC patients are two-fold: (1) Develop a core set of cognitive function, event related potential (ERP) measures from electroencephalogram (EEG), and resting-state functional magnetic resonance imaging (rsfMRI) measures to elucidate the relationship between impaired attentional control and EFN dysfunction and (2) Increase understanding of the link between neurocognitive impairment with concurrent symptom severity and impact on functioning. The investigators propose a longitudinal, prospective cohort pilot design to study post-operative CRC patients scheduled to begin adjuvant chemotherapy (Ctx+ group). Comparison groups will include post-operative CRC patients not receiving chemotherapy (Ctx- group) and healthy controls demographically matched to Ctx+ participants (HC group). All participants (N=60; 20 per group) will complete an additional 1-hour study visits at baseline and 24-weeks to collect rsfMRI measurements Ctx+ patients will complete baseline assessment after surgery but before starting chemotherapy, CTx- patients will complete baseline assessments 4-6 weeks after surgery and HC after matched and consented.

ELIGIBILITY:
Inclusion Criteria:

CRC adenocarcinoma patients:

* Stage II/IV patients receiving adjuvant CTX (Ctx+ group)
* Stage I/III patients not receiving CTX (Ctx- group)
* Normal or corrected to normal vision (corrected far visual acuity of 20/50 or better)

For demographically-matched healthy controls (HC group)

* Matched to patient receiving CTX on demographics: age (plus or minus 5 years, gender, race, menopausal status, and education (plus or minus 2 years)
* Normal or corrected-to-normal vision (corrected far visual acuity of 20/50 or better)

Exclusion Criteria:

CRC patients:

Cancer diagnosis/treatment in last 3 yrs. in addition to CRC (exceptionpatients with localized skin cancer) Prior chemotherapy within 1 year for CRC Cognitive impairment (MMSE score < 25) prior to baseline assessment

Demographically-matched healthy controls:

CRC cancer diagnosis All exclusion criteria for CRC patients.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CRC Diagnosis:
  Worse prognosis includes presentation with complete colon obstruction, perforation, T4 tumor fewer than 12 lymph nodes examined, elevated CEA levels pre-or post-surgery, positive margins, and peri-neural, lymphatic or venous invasion. Molecular markers also correlate with the aggressiveness of colon cancer.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Change from Trails A baseline at 12 weeks and 24 weeks (Specific Aim 1) | Change from baseline to 12 and 24 weeks
  Neurocognitive measure of processing speed; Completion time (milliseconds), where longer completion times are interpreted as slower processing speed
Change from Trails B baseline at 12 weeks and 24 weeks (Specific Aim 1) | Change from baseline to 12 weeks and 24 weeks
  Neurocognitive measure of executive functioning; Completion time (milliseconds) where larger differences in completion time are interpreted as slower executive functioning processes
Change from Symbol Digit Modalities baseline at 12 weeks and 24 weeks (Specific Aim 1) | Change from baseline to 12 weeks and 24 weeks
  Neurocognitive measure of psychomotor speed; Total correct complete, where greater number completed is interpreted as faster psychomotor speed
Change from Stroop baseline at 12 weeks and 24 weeks (Specific Aim 1) | Change from baseline to 12 weeks and 24 weeks
  Neurocognitive measure of inhibitory control; Total number completed, where greater number completed is interpreted as better inhibitory control.Interference scores are obtained to estimate inhibitory control, where more negative values are interpreted as lower inhibitory control (estimated by subtracting expected performance from observed performance in color-word condition)
Change from Auditory Verbal Learning Task baseline at 12 weeks and 24 weeks (Specific Aim 1) | Change from Baseline to 12 and 24 weeks
  Neurocognitive measure of verbal memory; Total number recalled (immediate), where greater number immediately recalled is interpreted as better verbal short-term memory. Total number recalled (delayed), where greater number recall following delay is interpreted as better verbal long-term memory
Change from Visual Search Performance baseline at 12 weeks and 24 weeks (Specific Aim IIa) | Change from baseline to 12 and 24 weeks
  Measure of Response time (milliseconds), where longer response times are interpreted as slower processing speed and lower inhibitory control.
Change from Change Detection Performance baseline at 12 weeks and 24 weeks (Specific Aim IIa) | Change from baseline to 12 and 24 weeks
  Measure of response accuracy, where larger response accuracies are interpreted as larger working memory capacity and higher inhibitory control.
Change from N2pc amplitude during visual search baseline at 12 weeks and 24 weeks (Specific Aim IIa) | Change from baseline to 12 and 24 weeks
  Measure of attentional control. Larger amplitudes are interpreted as more resources allocated towards stimulus selection and poor attentional control
Change from Contralateral delay activity (CDA) amplitude change during task performance baseline at 12 weeks and 24 weeks (Specific Aim IIa) | Change from baseline to 12 and 24 weeks
  Measure of working memory storage. Where larger amplitudes are interpreted as more resources allocated towards working memory storage.
Change from MRI white matter volume baseline at 12 weeks and 24 weeks (Specific Aim IIb) | Change from baseline to 6 months (only CTx+ group)
  Measure of white matter volume within executive function network
Change from MRI Grey matter volume baseline at 12 weeks and 24 weeks (Specific Aim IIb) | Change from baseline to 6 months (only CTx+ group)
  Measure of grey matter volume within executive function network
Change from Executive Functional Network functional connectivity baseline at 12 weeks and 24 weeks (Specific Aim IIb) | Change from baseline to 6 months (only CTx+ group)
  EFN function
Change from M.D. Anderson Symptom Inventory-Gastro-Intestinal (MDASI-GI) baseline at 12 weeks and 24 weeks(Specific Aim III) | Change from baseline to 12 weeks and 24 weeks
  Measures co-occurring symptom severity and interference with function
Change from Research And Development (RAND) Short Form-12 (SF-12) from baseline to 12 and 24 weeks (Specific Aim III) | Change from baseline to 12 weeks and 24 weeks
  Measures physical and mental functional status
Change from Functional Assessment of Cancer Therapy- Cognitive (FACT-COG) at baseline to 12 and 24 weeks (Specific Aim III) | Change from baseline to12 weeks and 24 weeks
  Self-perceives cognitive function
Change from Beck Depression Inventory (BDI) from baseline to 12 and 24 weeks (Specific Aim III) | Change from baseline to 12 and 24 weeks
  Assesses depressive symptoms

SECONDARY OUTCOMES:
Change from logMAR visual acuity baseline at 12 weeks and 24 weeks | Change from baseline to 12 and 24 weeks
  Measures visual acuity. Relatively lower logMAR values are interpreted as better visual acuity (estimated as log transformed estimate of visual acuity with respect to deviation from standard 20/20)
Change from logMAR contrast sensitivity baseline at 12 weeks and 24 weeks | Change from baseline to 12 and 24 weeks
  Measures contrast sensitivity. Relatively lower logMAR values are interpreted as better contrast sensitivity.
Change from Frequency Doubling Technology baseline at 12 weeks and 24 weeks | Change from baseline to 12 and 24 weeks
  Measures visual field loss. A binary (yes/no) variable where presence of visual field defect is coded as evidence of visual field loss
Change from Optical Coherence Tomography baseline at 12 weeks and 24 weeks | Change from baseline to 12 and 24 weeks
  Measure of retinal nerve fiber layer (RNFL) thickness

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Berger, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nerbaska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vardy JL, Dhillon HM, Pond GR, Rourke SB, Bekele T, Renton C, Dodd A, Zhang H, Beale P, Clarke S, Tannock IF. Cognitive Function in Patients With Colorectal Cancer Who Do and Do Not Receive Chemotherapy: A Prospective, Longitudinal, Controlled Study. J Clin Oncol. 2015 Dec 1;33(34):4085-92. doi: 10.1200/JCO.2015.63.0905. Epub 2015 Nov 2. PMID 26527785
- [Background] Vardy J, Dhillon HM, Pond GR, Rourke SB, Xu W, Dodd A, Renton C, Park A, Bekele T, Ringash J, Zhang H, Burkes R, Clarke SJ, Tannock IF. Cognitive function and fatigue after diagnosis of colorectal cancer. Ann Oncol. 2014 Dec;25(12):2404-2412. doi: 10.1093/annonc/mdu448. Epub 2014 Sep 11. PMID 25214544
- [Background] Myers JS. A comparison of the theory of unpleasant symptoms and the conceptual model of chemotherapy-related changes in cognitive function. Oncol Nurs Forum. 2009 Jan;36(1):E1-10. doi: 10.1188/09.ONF.E1-E10. PMID 19136326
- [Background] Von Ah D, Storey S, Jansen CE, Allen DH. Coping strategies and interventions for cognitive changes in patients with cancer. Semin Oncol Nurs. 2013 Nov;29(4):288-99. doi: 10.1016/j.soncn.2013.08.009. PMID 24183160
- [Background] Myers JS. Cancer- and chemotherapy-related cognitive changes: the patient experience. Semin Oncol Nurs. 2013 Nov;29(4):300-7. doi: 10.1016/j.soncn.2013.08.010. PMID 24183161
- [Background] Askren MK, Jung M, Berman MG, Zhang M, Therrien B, Peltier S, Ossher L, Hayes DF, Reuter-Lorenz PA, Cimprich B. Neuromarkers of fatigue and cognitive complaints following chemotherapy for breast cancer: a prospective fMRI investigation. Breast Cancer Res Treat. 2014 Sep;147(2):445-55. doi: 10.1007/s10549-014-3092-6. Epub 2014 Aug 21. PMID 25138546
- [Background] Jung MS, Zhang M, Askren MK, Berman MG, Peltier S, Hayes DF, Therrien B, Reuter-Lorenz PA, Cimprich B. Cognitive dysfunction and symptom burden in women treated for breast cancer: a prospective behavioral and fMRI analysis. Brain Imaging Behav. 2017 Feb;11(1):86-97. doi: 10.1007/s11682-016-9507-8. PMID 26809289
- [Background] Corbetta M, Shulman GL. Control of goal-directed and stimulus-driven attention in the brain. Nat Rev Neurosci. 2002 Mar;3(3):201-15. doi: 10.1038/nrn755. PMID 11994752
- [Background] Hopfinger JB, Buonocore MH, Mangun GR. The neural mechanisms of top-down attentional control. Nat Neurosci. 2000 Mar;3(3):284-91. doi: 10.1038/72999. PMID 10700262
- [Background] Wang L, Liu X, Guise KG, Knight RT, Ghajar J, Fan J. Effective connectivity of the fronto-parietal network during attentional control. J Cogn Neurosci. 2010 Mar;22(3):543-53. doi: 10.1162/jocn.2009.21210. PMID 19301995
- [Background] de Fockert J, Rees G, Frith C, Lavie N. Neural correlates of attentional capture in visual search. J Cogn Neurosci. 2004 Jun;16(5):751-9. doi: 10.1162/089892904970762. PMID 15200703
- [Background] Frick MA, Vachani CC, Hampshire MK, Bach C, Arnold-Korzeniowski K, Metz JM, Hill-Kayser CE. Survivorship after lower gastrointestinal cancer: Patient-reported outcomes and planning for care. Cancer. 2017 May 15;123(10):1860-1868. doi: 10.1002/cncr.30527. Epub 2017 Jan 5. PMID 28055110
- [Background] Arndt V, Merx H, Stegmaier C, Ziegler H, Brenner H. Quality of life in patients with colorectal cancer 1 year after diagnosis compared with the general population: a population-based study. J Clin Oncol. 2004 Dec 1;22(23):4829-36. doi: 10.1200/JCO.2004.02.018. PMID 15570086
- [Background] McCleary NJ, Odejide O, Szymonifka J, Ryan D, Hezel A, Meyerhardt JA. Safety and effectiveness of oxaliplatin-based chemotherapy regimens in adults 75 years and older with colorectal cancer. Clin Colorectal Cancer. 2013 Mar;12(1):62-9. doi: 10.1016/j.clcc.2012.09.001. Epub 2012 Oct 24. PMID 23102897
- [Background] Berger AM, Visovsky C, Hertzog M, Holtz S, Loberiza FR Jr. Usual and worst symptom severity and interference with function in breast cancer survivors. J Support Oncol. 2012 May-Jun;10(3):112-8. doi: 10.1016/j.suponc.2011.11.001. Epub 2012 Jan 24. PMID 22277573
- [Background] Berger AM, Grem JL, Visovsky C, Marunda HA, Yurkovich JM. Fatigue and other variables during adjuvant chemotherapy for colon and rectal cancer. Oncol Nurs Forum. 2010 Nov;37(6):E359-69. doi: 10.1188/10.ONF.E359-E369. PMID 21059569
- [Background] Berger AM, Mooney K, Alvarez-Perez A, Breitbart WS, Carpenter KM, Cella D, Cleeland C, Dotan E, Eisenberger MA, Escalante CP, Jacobsen PB, Jankowski C, LeBlanc T, Ligibel JA, Loggers ET, Mandrell B, Murphy BA, Palesh O, Pirl WF, Plaxe SC, Riba MB, Rugo HS, Salvador C, Wagner LI, Wagner-Johnston ND, Zachariah FJ, Bergman MA, Smith C; National comprehensive cancer network. Cancer-Related Fatigue, Version 2.2015. J Natl Compr Canc Netw. 2015 Aug;13(8):1012-39. doi: 10.6004/jnccn.2015.0122. PMID 26285247
- [Background] Berger AM, Mitchell SA, Jacobsen PB, Pirl WF. Screening, evaluation, and management of cancer-related fatigue: Ready for implementation to practice? CA Cancer J Clin. 2015 May-Jun;65(3):190-211. doi: 10.3322/caac.21268. Epub 2015 Mar 11. PMID 25760293
- [Background] Ahles TA, Root JC, Ryan EL. Cancer- and cancer treatment-associated cognitive change: an update on the state of the science. J Clin Oncol. 2012 Oct 20;30(30):3675-86. doi: 10.1200/JCO.2012.43.0116. Epub 2012 Sep 24. PMID 23008308
- [Background] Jim HS, Phillips KM, Chait S, Faul LA, Popa MA, Lee YH, Hussin MG, Jacobsen PB, Small BJ. Meta-analysis of cognitive functioning in breast cancer survivors previously treated with standard-dose chemotherapy. J Clin Oncol. 2012 Oct 10;30(29):3578-87. doi: 10.1200/JCO.2011.39.5640. Epub 2012 Aug 27. PMID 22927526
- [Background] Merriman JD, Von Ah D, Miaskowski C, Aouizerat BE. Proposed mechanisms for cancer- and treatment-related cognitive changes. Semin Oncol Nurs. 2013 Nov;29(4):260-9. doi: 10.1016/j.soncn.2013.08.006. PMID 24183157
- [Background] Du XL, Cai Y, Symanski E. Association between chemotherapy and cognitive impairments in a large cohort of patients with colorectal cancer. Int J Oncol. 2013 Jun;42(6):2123-33. doi: 10.3892/ijo.2013.1882. Epub 2013 Apr 4. PMID 23563930
- [Background] Lepage C, Smith AM, Moreau J, Barlow-Krelina E, Wallis N, Collins B, MacKenzie J, Scherling C. A prospective study of grey matter and cognitive function alterations in chemotherapy-treated breast cancer patients. Springerplus. 2014 Aug 19;3:444. doi: 10.1186/2193-1801-3-444. eCollection 2014. PMID 25184110
- [Background] Amidi A, Agerbaek M, Wu LM, Pedersen AD, Mehlsen M, Clausen CR, Demontis D, Borglum AD, Harboll A, Zachariae R. Changes in cognitive functions and cerebral grey matter and their associations with inflammatory markers, endocrine markers, and APOE genotypes in testicular cancer patients undergoing treatment. Brain Imaging Behav. 2017 Jun;11(3):769-783. doi: 10.1007/s11682-016-9552-3. PMID 27240852
- [Background] McDonald BC, Conroy SK, Ahles TA, West JD, Saykin AJ. Alterations in brain activation during working memory processing associated with breast cancer and treatment: a prospective functional magnetic resonance imaging study. J Clin Oncol. 2012 Jul 10;30(20):2500-8. doi: 10.1200/JCO.2011.38.5674. Epub 2012 Jun 4. PMID 22665542
- [Background] McDonald BC, Conroy SK, Ahles TA, West JD, Saykin AJ. Gray matter reduction associated with systemic chemotherapy for breast cancer: a prospective MRI study. Breast Cancer Res Treat. 2010 Oct;123(3):819-28. doi: 10.1007/s10549-010-1088-4. Epub 2010 Aug 6. PMID 20690040
- [Background] Deprez S, Amant F, Smeets A, Peeters R, Leemans A, Van Hecke W, Verhoeven JS, Christiaens MR, Vandenberghe J, Vandenbulcke M, Sunaert S. Longitudinal assessment of chemotherapy-induced structural changes in cerebral white matter and its correlation with impaired cognitive functioning. J Clin Oncol. 2012 Jan 20;30(3):274-81. doi: 10.1200/JCO.2011.36.8571. Epub 2011 Dec 19. PMID 22184379
- [Background] Kam JWY, Brenner CA, Handy TC, Boyd LA, Liu-Ambrose T, Lim HJ, Hayden S, Campbell KL. Sustained attention abnormalities in breast cancer survivors with cognitive deficits post chemotherapy: An electrophysiological study. Clin Neurophysiol. 2016 Jan;127(1):369-378. doi: 10.1016/j.clinph.2015.03.007. Epub 2015 Mar 21. PMID 25868929
- [Background] Kreukels BP, van Dam FS, Ridderinkhof KR, Boogerd W, Schagen SB. Persistent neurocognitive problems after adjuvant chemotherapy for breast cancer. Clin Breast Cancer. 2008 Feb;8(1):80-7. doi: 10.3816/CBC.2008.n.006. PMID 18501062
- [Background] Kreukels BP, Schagen SB, Ridderinkhof KR, Boogerd W, Hamburger HL, van Dam FS. Electrophysiological correlates of information processing in breast-cancer patients treated with adjuvant chemotherapy. Breast Cancer Res Treat. 2005 Nov;94(1):53-61. doi: 10.1007/s10549-005-7093-3. PMID 16175317
- [Background] Kreukels BP, Schagen SB, Ridderinkhof KR, Boogerd W, Hamburger HL, Muller MJ, van Dam FS. Effects of high-dose and conventional-dose adjuvant chemotherapy on long-term cognitive sequelae in patients with breast cancer: an electrophysiologic study. Clin Breast Cancer. 2006 Apr;7(1):67-78. doi: 10.3816/CBC.2006.n.015. PMID 16764746
- [Background] Bender CM, Thelen BD. Cancer and cognitive changes: the complexity of the problem. Semin Oncol Nurs. 2013 Nov;29(4):232-7. doi: 10.1016/j.soncn.2013.08.003. PMID 24183154
- [Background] Von Ah D. Cognitive changes associated with cancer and cancer treatment: state of the science. Clin J Oncol Nurs. 2015 Feb;19(1):47-56. doi: 10.1188/15.CJON.19-01AP. PMID 25689649
- [Background] Hedayati E, Alinaghizadeh H, Schedin A, Nyman H, Albertsson M. Effects of adjuvant treatment on cognitive function in women with early breast cancer. Eur J Oncol Nurs. 2012 Jul;16(3):315-22. doi: 10.1016/j.ejon.2011.07.006. Epub 2011 Sep 9. PMID 21908235
- [Background] Quesnel C, Savard J, Ivers H. Cognitive impairments associated with breast cancer treatments: results from a longitudinal study. Breast Cancer Res Treat. 2009 Jul;116(1):113-23. doi: 10.1007/s10549-008-0114-2. Epub 2008 Jul 16. PMID 18629633
- [Background] Shilling V, Jenkins V, Morris R, Deutsch G, Bloomfield D. The effects of adjuvant chemotherapy on cognition in women with breast cancer--preliminary results of an observational longitudinal study. Breast. 2005 Apr;14(2):142-50. doi: 10.1016/j.breast.2004.10.004. PMID 15767184
- [Background] Stewart A, Collins B, Mackenzie J, Tomiak E, Verma S, Bielajew C. The cognitive effects of adjuvant chemotherapy in early stage breast cancer: a prospective study. Psychooncology. 2008 Feb;17(2):122-30. doi: 10.1002/pon.1210. PMID 17518411
- [Background] Tager FA, McKinley PS, Schnabel FR, El-Tamer M, Cheung YK, Fang Y, Golden CR, Frosch ME, Habif U, Mulligan MM, Chen IS, Hershman DL. The cognitive effects of chemotherapy in post-menopausal breast cancer patients: a controlled longitudinal study. Breast Cancer Res Treat. 2010 Aug;123(1):25-34. doi: 10.1007/s10549-009-0606-8. Epub 2009 Nov 6. PMID 19894112
- [Background] Collins B, Mackenzie J, Stewart A, Bielajew C, Verma S. Cognitive effects of hormonal therapy in early stage breast cancer patients: a prospective study. Psychooncology. 2009 Aug;18(8):811-21. doi: 10.1002/pon.1453. PMID 19085975
- [Background] Wefel JS, Vidrine DJ, Marani SK, Swartz RJ, Veramonti TL, Meyers CA, Hoekstra HJ, Hoekstra-Weebers JE, Gritz ER. A prospective study of cognitive function in men with non-seminomatous germ cell tumors. Psychooncology. 2014 Jun;23(6):626-33. doi: 10.1002/pon.3453. Epub 2013 Dec 16. PMID 24339329
- [Background] Cruzado JA, Lopez-Santiago S, Martinez-Marin V, Jose-Moreno G, Custodio AB, Feliu J. Longitudinal study of cognitive dysfunctions induced by adjuvant chemotherapy in colon cancer patients. Support Care Cancer. 2014 Jul;22(7):1815-23. doi: 10.1007/s00520-014-2147-x. Epub 2014 Feb 18. PMID 24535240
- [Background] Collins B, MacKenzie J, Tasca GA, Scherling C, Smith A. Cognitive effects of chemotherapy in breast cancer patients: a dose-response study. Psychooncology. 2013 Jul;22(7):1517-27. doi: 10.1002/pon.3163. Epub 2012 Aug 30. PMID 22936651
- [Background] Deprez S, Amant F, Yigit R, Porke K, Verhoeven J, Van den Stock J, Smeets A, Christiaens MR, Leemans A, Van Hecke W, Vandenberghe J, Vandenbulcke M, Sunaert S. Chemotherapy-induced structural changes in cerebral white matter and its correlation with impaired cognitive functioning in breast cancer patients. Hum Brain Mapp. 2011 Mar;32(3):480-93. doi: 10.1002/hbm.21033. PMID 20725909
- [Background] Ahles TA, Saykin AJ, McDonald BC, Li Y, Furstenberg CT, Hanscom BS, Mulrooney TJ, Schwartz GN, Kaufman PA. Longitudinal assessment of cognitive changes associated with adjuvant treatment for breast cancer: impact of age and cognitive reserve. J Clin Oncol. 2010 Oct 10;28(29):4434-40. doi: 10.1200/JCO.2009.27.0827. Epub 2010 Sep 13. PMID 20837957
- [Background] Jenkins V, Thwaites R, Cercignani M, Sacre S, Harrison N, Whiteley-Jones H, Mullen L, Chamberlain G, Davies K, Zammit C, Matthews L, Harder H. A feasibility study exploring the role of pre-operative assessment when examining the mechanism of 'chemo-brain' in breast cancer patients. Springerplus. 2016 Mar 31;5:390. doi: 10.1186/s40064-016-2030-y. eCollection 2016. PMID 27047716
- [Background] Kreukels BPC, Hamburger HL, de Ruiter MB, van Dam FSAM, Ridderinkhof KR, Boogerd W, Schagen SB. ERP amplitude and latency in breast cancer survivors treated with adjuvant chemotherapy. Clin Neurophysiol. 2008 Mar;119(3):533-541. doi: 10.1016/j.clinph.2007.11.011. PMID 18164658
- [Background] Luck SJ, Hillyard SA. Electrophysiological correlates of feature analysis during visual search. Psychophysiology. 1994 May;31(3):291-308. doi: 10.1111/j.1469-8986.1994.tb02218.x. PMID 8008793
- [Background] Vogel EK, Machizawa MG. Neural activity predicts individual differences in visual working memory capacity. Nature. 2004 Apr 15;428(6984):748-51. doi: 10.1038/nature02447. PMID 15085132
- [Background] Painter DR, Dux PE, Mattingley JB. Distinct roles of the intraparietal sulcus and temporoparietal junction in attentional capture from distractor features: An individual differences approach. Neuropsychologia. 2015 Jul;74:50-62. doi: 10.1016/j.neuropsychologia.2015.02.029. Epub 2015 Feb 24. PMID 25724234
- [Background] Harris AM, Dux PE, Jones CN, Mattingley JB. Distinct roles of theta and alpha oscillations in the involuntary capture of goal-directed attention. Neuroimage. 2017 May 15;152:171-183. doi: 10.1016/j.neuroimage.2017.03.008. Epub 2017 Mar 6. PMID 28274832
- [Background] Vogel EK, McCollough AW, Machizawa MG. Neural measures reveal individual differences in controlling access to working memory. Nature. 2005 Nov 24;438(7067):500-3. doi: 10.1038/nature04171. PMID 16306992
- [Background] Lopez Zunini RA, Scherling C, Wallis N, Collins B, MacKenzie J, Bielajew C, Smith AM. Differences in verbal memory retrieval in breast cancer chemotherapy patients compared to healthy controls: a prospective fMRI study. Brain Imaging Behav. 2013 Dec;7(4):460-77. doi: 10.1007/s11682-012-9213-0. PMID 23242968
- [Background] Schrepf A, Lutgendorf SK, Pyter LM. Pre-treatment effects of peripheral tumors on brain and behavior: neuroinflammatory mechanisms in humans and rodents. Brain Behav Immun. 2015 Oct;49:1-17. doi: 10.1016/j.bbi.2015.04.010. Epub 2015 May 6. PMID 25958011
- [Background] Bower JE. Cancer-related fatigue--mechanisms, risk factors, and treatments. Nat Rev Clin Oncol. 2014 Oct;11(10):597-609. doi: 10.1038/nrclinonc.2014.127. Epub 2014 Aug 12. PMID 25113839
- [Background] Cashdollar N, Fukuda K, Bocklage A, Aurtenetxe S, Vogel EK, Gazzaley A. Prolonged disengagement from attentional capture in normal aging. Psychol Aging. 2013 Mar;28(1):77-86. doi: 10.1037/a0029899. Epub 2012 Oct 15. PMID 23066799
- [Background] Jost K, Bryck RL, Vogel EK, Mayr U. Are old adults just like low working memory young adults? Filtering efficiency and age differences in visual working memory. Cereb Cortex. 2011 May;21(5):1147-54. doi: 10.1093/cercor/bhq185. Epub 2010 Sep 30. PMID 20884722
- [Background] Vakoc BJ, Fukumura D, Jain RK, Bouma BE. Cancer imaging by optical coherence tomography: preclinical progress and clinical potential. Nat Rev Cancer. 2012 Apr 5;12(5):363-8. doi: 10.1038/nrc3235. PMID 22475930
- [Background] Wang XS, Williams LA, Eng C, Mendoza TR, Shah NA, Kirkendoll KJ, Shah PK, Trask PC, Palos GR, Cleeland CS. Validation and application of a module of the M. D. Anderson Symptom Inventory for measuring multiple symptoms in patients with gastrointestinal cancer (the MDASI-GI). Cancer. 2010 Apr 15;116(8):2053-63. doi: 10.1002/cncr.24920. PMID 20166216
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Lai JS, Butt Z, Wagner L, Sweet JJ, Beaumont JL, Vardy J, Jacobsen PB, Shapiro PJ, Jacobs SR, Cella D. Evaluating the dimensionality of perceived cognitive function. J Pain Symptom Manage. 2009 Jun;37(6):982-95. doi: 10.1016/j.jpainsymman.2008.07.012. PMID 19500722
- [Background] Smith S, Jenkinson M, Beckmann C, Miller K, Woolrich M. Meaningful design and contrast estimability in FMRI. Neuroimage. 2007 Jan 1;34(1):127-36. doi: 10.1016/j.neuroimage.2006.09.019. Epub 2006 Oct 27. PMID 17070706
- [Background] Desmond JE, Glover GH. Estimating sample size in functional MRI (fMRI) neuroimaging studies: statistical power analyses. J Neurosci Methods. 2002 Aug 30;118(2):115-28. doi: 10.1016/s0165-0270(02)00121-8. PMID 12204303
- [Background] Birn RM, Molloy EK, Patriat R, Parker T, Meier TB, Kirk GR, Nair VA, Meyerand ME, Prabhakaran V. The effect of scan length on the reliability of resting-state fMRI connectivity estimates. Neuroimage. 2013 Dec;83:550-8. doi: 10.1016/j.neuroimage.2013.05.099. Epub 2013 Jun 6. PMID 23747458
- [Background] Pajula J, Tohka J. How Many Is Enough? Effect of Sample Size in Inter-Subject Correlation Analysis of fMRI. Comput Intell Neurosci. 2016;2016:2094601. doi: 10.1155/2016/2094601. Epub 2016 Jan 13. PMID 26884746
- [Derived] Berger AM, Grem J, Garlinghouse M, Lyden E, Schmid K. Neurocognitive function and quality-of-life in patients with colorectal cancer. Eur J Oncol Nurs. 2023 Jun;64:102304. doi: 10.1016/j.ejon.2023.102304. Epub 2023 Mar 24. PMID 37137248